CLINICAL TRIAL: NCT04175535
Title: The Comparative Study of Full-Endoscopic Cervical Posterior Discectomy and Anterior Cervical Decompression and Fusion for the Operation of Soft Cervical Disc Herniation.
Brief Title: The Comparative Study of Full-Endoscopic Cervical Posterior Discectomy and Anterior Cervical Decompression and Fusion
Acronym: PPECD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: zeyy1985811
Record Dates: First submitted 2019-10-17; First posted 2019-11-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: M-JOA Score
Keywords: cervical disc herniation; endoscope; posterior; minimally invasive spine surgery
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were unaware of the grouping process. The surgeons were unaware of the grouping process. The follow-up recorders were unaware of the grouping process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Other): PPECD was performed in the experimental group
  Interventions: Procedure: Percutaneous Posterior Endoscopic Cervical Discectomy
- control group (Other): ACDF was performed in the control group
  Interventions: Procedure: Anterior cervical decompression and fusion

INTERVENTIONS:
Procedure: Percutaneous Posterior Endoscopic Cervical Discectomy — The most common alternative in the case of soft cervical disc herniations.
  Arms: The experimental group
Procedure: Anterior cervical decompression and fusion — The standard procedure for operation of cervical disc herniations.
  Arms: control group

SUMMARY:
Anterior cervical decompression and fusion is the standard procedure for operation of cervical disc herniations. Mobility-preserving Full-Endoscopic Cervical Posterior discectomy is the most common alternative in the case of soft localization of the pathology. Endoscopic techniques are considered standard in many areas, since they may offer advantages in surgical technique and rehabilitation. These days, all disc herniations can be operated in full-endoscopic technique. With the full-endoscopic posterior cervical discectomy a procedures is available for cervical disc operations.

DETAILED DESCRIPTION:
Investigators conducted a differential, randomized, 1:1, double-blind clinical control trial to compare the clinical effect, safety and feasibility of Full-Endoscopic Cervical Posterior discectomy and Anterior cervical decompression and fusion. The study was conducted in three centers at the same time, including the Second Affiliated Hospital of Zhejiang University Medical College, Zhejiang Provincial People's Hospital and Ningbo University Medical College Affiliated Hospital. This study is expected to include 308 patients with single level soft cervical disc herniation.Participants were randomly assigned to different groups for corresponding surgical intervention after complete preoperative evaluation.Participants received a standard 5-year follow-up procedure

ELIGIBILITY:
Inclusion Criteria:

1. Single cervical intervertebral dis herniation wih symptoms of radicular pain or spinal cord compression ; 2) the herniated lesions had no obvious calcification; 3) conservative treatment fails ; 4) mild myelopathy (Nurick grade 3 or blow. (6) patients agree to participate in this study.

Exclusion Criteria:

1. cervical segmental instability or deformity (cervical spondylolisthesis or Cobb Angle greater than 25°); 2) multisegmental lesions (≥2); 3) tumor, infection or other unknown space occupying in cervical vertebra; 4) surgical history of the target segment; 5) severe myelopathy (Nurick grade 4 or above); 6) the patients were not suitable for surgery, had poor medical management or did not agree to participate in this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement rate | Follow up for 5 years
  M-JOA Scoring

SECONDARY OUTCOMES:
Basic information of participants | Follow up for 5 years
  Age in year, gender in male or female, occupation
Basic information of participants | Follow up for 5 years
  weight and height will be combined to report BMI in kg/m^2
Imaging examination | Follow up for 5 years
  Cervical cobb angle change i
Pain Assessment | Follow up for 5 years
  VAS Score
Operation duration | intraoperative
  Operation duration in minute
Amount of bleeding during operation | Follow up for 5 years
  Amount of bleeding during operation in milliliter

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No